CLINICAL TRIAL: NCT06250647
Title: Effect of Dietary Intervention With a High Intake of Vitamin K on Insulin, Osteocalcin, Leptin, Vitamin K Serum Levels and Cardiovascular Risk in Young Adults With and Without Overweight or Obesity.
Brief Title: High Vitamin K Intake Diet Intervention Effect on Cardiovascular Risk Percentage in Young Adults
Acronym: VKDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CI-04720; 20-18 (Other: Universidad de Guadalajara)
Record Dates: First submitted 2023-11-27; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Overweight and Obesity
Keywords: Vitamin K; diet intervention; Cardiovascular disease; overweight and obesity; young adults
MeSH Terms: conditions — Overweight; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VK INTERVENTION (Experimental): administration of a menu diet containing 500mcg of vitamin K (in the food selected) durinf 6 weeks.
  Interventions: Other: vitamin K diet
- DIETARY RECOMMENDATIONS (No Intervention): No menu administration but only recommendations for correct diet.

INTERVENTIONS:
Other: vitamin K diet — 500mcg of Vitamin K intake provided by the selection of vitamin k rich foods in the menu.
  Arms: VK INTERVENTION

SUMMARY:
The goal of this clinical trial is to compare the effect of a high vitamin K diet intervention on vitamin K, insulin, osteocalcin serum levels and the cardiovascular risk percentage in normal weight and overweight or obese young adults. The main questions it aims to answer are: • Does a diet intervention containing 500mcg of vitamin K increases serum vitamin K levels? • Are vitamin K serum levels after the 500mcg of vitamin K diet intervention associated with insulin and osteocalcin serum levels or the cardiovascular risk percentage in normal weight and overweight or obese young adults? Participants will have to follow a diet intervention that contains 500mcg of vitamin K, given as a cyclic menu for 6 weeks. Also, participants will have to assist weekly to nutritional monitoring and to report any situation they observed regarding the intervention during this study. Researchers will compare normal weight and overweight or obese groups with diet intervention with normal weight and overweight or obese groups without diet intervention and only dietetic recommendations to see if vitamin K serum levels, insulin, osteocalcin and the cardiovascular risk percentage improve after the 6 weeks diet intervention.

ELIGIBILITY:
Inclusion Criteria:

* young adults
* acceptation for participate
* acceptation to asist to monitoring sessions
* sign information consent

Exclusion Criteria:

* under other dietetic intervention
* under medications that interfere with vitamin K or diminish its absorbtion
* vitamin E or A intake supplements
* previous diagnose of metabolic syndrome, diabetes mellitus, hypertension, cancer or dyslipidemia.
* chronic alcohol intake
* some medical or health situation that impedes the following of the program

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-02-06 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
vitamin K serum levels | basal and after 6 weeks of diet intervention
  ng/mL
Cardiovascular Risk Percentage | basal and after 6 weeks of diet intervention
  percentage (%)
insulin serum levels | basal and after 6 weeks of diet intervention
  mcUI/L

SECONDARY OUTCOMES:
Osteocalcin | basal and after 6 weeks of diet intervention
  ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Iris M Llamas-Covarrubias, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Centro Universitario de Ciencias de la Salud, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication
Access Criteria: IPD will be shared by email request after the request review by the main researcher

REFERENCES:
- [Background] Chen HG, Sheng LT, Zhang YB, Cao AL, Lai YW, Kunutsor SK, Jiang L, Pan A. Association of vitamin K with cardiovascular events and all-cause mortality: a systematic review and meta-analysis. Eur J Nutr. 2019 Sep;58(6):2191-2205. doi: 10.1007/s00394-019-01998-3. Epub 2019 May 22. PMID 31119401
- [Background] Simes DC, Viegas CSB, Araujo N, Marreiros C. Vitamin K as a Diet Supplement with Impact in Human Health: Current Evidence in Age-Related Diseases. Nutrients. 2020 Jan 3;12(1):138. doi: 10.3390/nu12010138. PMID 31947821
- [Background] Vera-Remartinez EJ, Lazaro Monge R, Granero Chinesta S, Sanchez-Alcon Rodriguez D, Planelles Ramos MV. [Cardiovascular risk factors in young adults of a penitentiary center]. Rev Esp Salud Publica. 2018 Jul 6;92:e201807037. Spanish. PMID 29978853
- [Background] Shea MK, Booth SL, Weiner DE, Brinkley TE, Kanaya AM, Murphy RA, Simonsick EM, Wassel CL, Vermeer C, Kritchevsky SB; Health ABC Study. Circulating Vitamin K Is Inversely Associated with Incident Cardiovascular Disease Risk among Those Treated for Hypertension in the Health, Aging, and Body Composition Study (Health ABC). J Nutr. 2017 May;147(5):888-895. doi: 10.3945/jn.117.249375. Epub 2017 Mar 29. PMID 28356433
- [Background] Yoshida M, Booth SL, Meigs JB, Saltzman E, Jacques PF. Phylloquinone intake, insulin sensitivity, and glycemic status in men and women. Am J Clin Nutr. 2008 Jul;88(1):210-5. doi: 10.1093/ajcn/88.1.210. PMID 18614743
- [Background] Al-Suhaimi EA, Al-Jafary MA. Endocrine roles of vitamin K-dependent- osteocalcin in the relation between bone metabolism and metabolic disorders. Rev Endocr Metab Disord. 2020 Mar;21(1):117-125. doi: 10.1007/s11154-019-09517-9. PMID 31761961
- [Result] Gaona-Pineda EB, Martinez-Tapia B, Arango-Angarita A, Valenzuela-Bravo D, Gomez-Acosta LM, Shamah-Levy T, Rodriguez-Ramirez S. [Food groups consumption and sociodemographic characteristics in Mexican population]. Salud Publica Mex. 2018 May-Jun;60(3):272-282. doi: 10.21149/8803. Spanish. PMID 29746744

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT06250647/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT06250647/ICF_001.pdf